CLINICAL TRIAL: NCT02091310
Title: A Two-part Phase I Study Composed of a Randomized, Double-blind, 4-parallel Group Study to Evaluate the Effect of Multiple Oral Doses of GFT505 on the QT/QTc Interval Compared to Placebo With Moxifloxacin (400 mg in Single Oral Dose) as a Positive Control, in Healthy Male and Female Volunteers, Preceded by a Double-blind, Placebo-controlled, Safety, Tolerability and Pharmacokinetic Study in Healthy Male Volunteers in Order to Define the Supra-therapeutic GFT505 Dose in a Multiple Dosing Regimen.
Brief Title: Phase I Study to Evaluate the Effect of GFT505 on QT/QTc Interval in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genfit (Industry)
Collaborators: Eurofins Optimed (Industry); CardiaBase (Other); PhinC Development (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GFT505-113-9; 2013-005154-30 (EudraCT Number)
Record Dates: First submitted 2014-03-14; First posted 2014-03-19 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Healthy Volunteers
Keywords: GFT505; TQT; QT/QTc; Pharmacokinetic; Healthy subjects; Moxifloxacin
MeSH Terms: interventions — 2-(2,6-dimethyl-4-(3-(4-(methylthio)phenyl)-3-oxo-1-propenyl)phenoxyl)-2-methylpropanoic acid; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- Placebo (Study Part I) (Placebo Comparator): Hard gelatin capsules, oral administration, 5 or 6 capsules per day before breakfast with a glass of water
  Interventions: Drug: Placebo
- GFT505 300 mg (Study Part I) (Experimental): Hard gelatin capsules dosed at 60mg, oral administration, 5 capsules per day before breakfast with a glass of water
  Interventions: Drug: GFT505
- GFT505 360 mg (Study Part I) (Experimental): Hard gelatin capsules dosed at 60mg, oral administration, 6 capsules per day before breakfast with a glass of water
  Interventions: Drug: GFT505
- Placebo (Study Part II) (Placebo Comparator): Hard gelatin capsules, oral administration, 4 to 6 capsules per day before breakfast with a glass of water
  Interventions: Drug: Placebo
- GFT505 120 mg (Study Part II) (Experimental): Hard gelatin capsules dosed at 60mg, oral administration, 2 capsules per day plus 2 to 4 capsules of placebo per day before breakfast with a glass of water
  Interventions: Drug: GFT505
- GFT505 xx mg (Study Part II) (Experimental): Supra-therapeutic dose: hard gelatin capsules dosed at 60mg, oral administration, 4 to 6 capsules per day before breakfast with a glass of water
  Interventions: Drug: GFT505
- Moxifloxacin 400 mg (Study Part II) (Active Comparator): On days 1 to 13, 4 to 6 placebo capsules per day, then one 400 mg moxifloxacin tablet (Izilox®, Bayer Pharmaceuticals Corporation) administered orally on Day 14
  Interventions: Drug: Moxifloxacin 400 mg

INTERVENTIONS:
Drug: Placebo
  Arms: Placebo (Study Part I); Placebo (Study Part II)
Drug: GFT505
  Arms: GFT505 120 mg (Study Part II); GFT505 300 mg (Study Part I); GFT505 360 mg (Study Part I); GFT505 xx mg (Study Part II)
Drug: Moxifloxacin 400 mg
  Arms: Moxifloxacin 400 mg (Study Part II)

SUMMARY:
In accordance with International Conference on Harmonisation (ICH) E14 guidelines, this Phase I thorough QT (TQT) study will assess the arrhythmogenic potential of GFT505, by evaluating its effect on QT/QTc prolongation in healthy male and female subjects. According to the guidelines, such studies should typically be performed at the expected therapeutic dose and a supra-therapeutic dose that is 3-4-fold higher than the therapeutic dose.

GFT505 has previously been tested at 240 mg/d in 14-day multiple administration to healthy overweight subjects (study GFT505-111-7), and both safety and tolerability were very good. However, this dose corresponds to only 2-fold the expected therapeutic dose of 120 mg/d. Therefore, the current TQT study will be preceded by a multiple ascending dose study in which the safety and tolerability of 2 dose levels of GFT505 (300 and 360 mg) corresponding to 2.5 and 3 times the expected therapeutic dose will be evaluated. The highest dose level for which safety and tolerability are considered satisfactory will be the supra-therapeutic dose used in the TQT study.

DETAILED DESCRIPTION:
The present trial is split into two successive parts:

* Study Part I is a double-blind, randomized, placebo-controlled study designed to obtain safety, tolerability and pharmacokinetic (PK) data after 14-day multiple oral administrations of once-daily increasing doses of GFT505 (300 and 360 mg) in healthy male subjects. The starting dose of 300 mg/day has been selected on the basis of the results of previous clinical trials and corresponds to the highest dose given in healthy subjects according to a single dose regimen (study GFT505-111-7). A total of 24 male subjects will be included, 12 for each cohort (a cohort corresponding to a dose level). In each cohort, 9 subjects will receive GFT505 and 3 will receive placebo. A Safety Review Committee (SRC) will have a formal meeting after full completion of at least 10 out of 12 subjects of each dose level to review under blinded conditions all safety data and to conclude on the safety and tolerability of a given dose level. Between the first and the second dose level, the SRC will give its agreement on the dose escalation, and at completion of the second level the SRC will define the supra-therapeutic dose to be administered in Study Part II.
* Study Part II will be a parallel group, randomized, placebo-controlled study, with stratification by gender. The study is designed to investigate the potential impact of 14-day multiple oral administrations of once-daily GFT505 on QT/QTc prolongation under conditions of maximal GFT505 exposure, i.e. by administering the expected therapeutic dose of 120 mg/d and a supra-therapeutic dose (defined according to the results of Study Part I), to healthy male and female subjects. A single oral dose of 400 mg moxifloxacin will be used as a positive control in order to document the sensitivity of the experimental conditions. The study treatment administration will be double-blind for placebo and GFT505 and open for moxifloxacin. The ECG readings will be performed under blinded conditions. A preliminary sample size of 128 subjects to have at least 124 evaluable subjects has been fixed by formal justification on a theoretical basis. ECG data collected during Study Part I will support a formal determination using observed data and thus will lead to a final sample size. In all cases, it is anticipated that the sample size could not be less than 124 evaluable subjects. Each gender will represent at least 40% of the study population. Both sub-groups will be balanced between the 4 treatment groups.

ELIGIBILITY:
Inclusion Criteria:

Part I:

* Healthy males aged 18 to 45 years inclusive
* Body Mass Index (BMI) ≥ 18 ≤ 30 kg/m²
* No clinically relevant abnormalities in blood pressure (BP) or heart rate (HR)
* No clinically relevant abnormalities in 12-lead ECG results

Part II:

* Healthy males and females aged 18 to 45 years inclusive
* For female subjects of childbearing potential, use of double contraception method
* Body Mass Index (BMI) ≥ 18 ≤ 30 kg/m²
* No clinically relevant abnormalities in blood pressure (BP) or heart rate (HR)
* No clinically relevant abnormalities in 12-lead ECG results

Exclusion Criteria:

Part I:

* Evidence of clinically relevant cardiovascular, renal, hepatic, hematological, gastrointestinal, pulmonary, metabolic-endocrine, neurological, urogenital or psychiatric diseases
* A history of risk factors for "Torsades de Pointe" (e.g., heart failure, hypokalemia, family history of Long QT Syndrome)
* Any condition requiring regular concomitant medication, including herbal products and over-the-counter (OTC) medication or predicted need of any concomitant medication during the study
* Current drug or alcohol abuse [including regular alcohol drinking of more than 21 units per week (1 unit = 4 cL spirits or equivalent)] or a history of drug or alcohol abuse within 1 year before screening
* Current use of nicotine containing products, i.e., more than 5 cigarettes or equivalent/day and the inability to stop using nicotine containing products during confinement in the clinical center
* Use of caffeine containing beverages exceeding 500 mg caffeine/day (5 cups of coffee) and the inability to refrain from the use of caffeine containing beverages during confinement in the clinical center
* Blood donation or loss of significant amount of blood within 2 months prior to the first dosing
* Any other condition that in the opinion of the Investigator would interfere with the evaluation of the results or constitute a health risk for the subject.

Part II:

* Evidence of clinically relevant cardiovascular, renal, hepatic, hematological, gastrointestinal, pulmonary, metabolic-endocrine, neurological, urogenital or psychiatric diseases
* A history of risk factors for "Torsades de Pointe" (e.g., heart failure, hypokalemia, family history of Long QT Syndrome)
* The use of concomitant medications that prolong the QT/QTc interval
* Any condition requiring regular concomitant medication, including herbal products and over-the-counter (OTC) medication or predicted need of any concomitant medication during the study
* Current drug or alcohol abuse [including regular alcohol drinking of more than 21 units (for male) or 14 units (for female) (1 unit = 4 cL spirits or equivalent)] or a history of drug or alcohol abuse within 1 year before screening
* Current use of nicotine containing products, i.e., more than 5 cigarettes or equivalent/day and the inability to stop using nicotine containing products during confinement in the clinical center
* Use of caffeine containing beverages exceeding 500 mg caffeine/day (5 cups of coffee) and the inability to refrain from the use of caffeine containing beverages during confinement in the clinical center
* Blood donation or loss of significant amount of blood within 2 months prior to the first dosing
* For women: Positive pregnancy test at screening or on Day -2; Pregnancy or trying to become pregnant; Breastfeeding
* Any other condition that in the opinion of the Investigator would interfere with the evaluation of the results or constitute a health risk for the subject.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2014-02; Primary Completion 2014-12 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Safety parameters such as adverse event monitoring, vital signs, ECG, and clinical laboratory tests (Study Part I) | 14 days
  To evaluate the safety and tolerability of two dose levels of GFT505 (300 and 360 mg), after multiple dose administration once daily for 14 days in male healthy subjects in order to determine the supra-therapeutic dose to be administered in Study Part II.
Effect on QTcF compared to placebo (Study Part II) | 14 days
  To evaluate the impact on QTcF of two dose levels (one therapeutic and one supra-therapeutic according to ICH E14) of GFT505, after multiple dose administration once daily for 14 days in healthy male and female subjects compared to placebo and a positive control.

SECONDARY OUTCOMES:
Pharmacokinetic parameters including Cmax, Tmax, AUCt (Study Part I) | 14 days
  To determine the PK parameters of GFT505 and GFT1007 after multiple dose administration once daily for 14 days in male subjects.
Safety parameters such as adverse event monitoring, vital signs, ECG, and clinical laboratory tests (Study Part II) | 14 days
  To evaluate the safety and tolerability of GFT505 in healthy male and female subjects after multiple dose administration of a therapeutic dose and a supra-therapeutic dose
Effect on QTcB compared to placebo (Study Part II) | 14 days
  To evaluate the impact on QTcB of two dose levels (one therapeutic and one supra-therapeutic according to ICH E14) of GFT505, after multiple dose administration once daily for 14 days in healthy male and female subjects compared to placebo and a positive control.

CONTACTS AND LOCATIONS:
Overall Officials: Rémy Hanf, PhD, Study Director — Genfit
Locations (1):
- Eurofins Optimed, Gières, France